CLINICAL TRIAL: NCT06797284
Title: The Impact of Light, Electrical, and Magnetic Neuroregulation Interventions on Sleep-wake Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chun-Feng Liu, professor, Second Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LK2024002
Record Dates: First submitted 2024-09-17; First posted 2025-01-28 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Insomnia Chronic; Narcolepsy; REM Sleep Behavior Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Narcolepsy; REM Sleep Behavior Disorder | interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation; Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Experimental): transcranial magnetic stimulation or transcranial direct current stimulation or daytime timed bright light exposure
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — repetitive transcranial magnetic stimulation, or transcranial direct current stimulation, or daytime timed bright light exposure
  Other Names: Transcranial Electrical Stimulation; light therapy

SUMMARY:
Carry out precise and effective neuromodulation interventions, and develop new neuromodulation technologies for sleep disorders. Use phototherapy, transcranial electrical/magnetic stimulation and other therapies to conduct self-controlled intervention studies on insomnia, narcolepsy, and rapid eye movement sleep behavior disorder .

ELIGIBILITY:
Inclusion Criteria:

- Patients with insomnia, narcolepsy,and RBD that have been clearly diagnosed by specialists should sign the informed consent form.

Exclusion Criteria:

1. Patients with major neurological diseases such as multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumors, progressive supranuclear palsy, epilepsy, subdural hematoma, multiple sclerosis, or those who have sustained neurological dysfunction or known structural brain abnormalities after significant head trauma are excluded.
2. A history of major depressive disorder or bipolar disorder within the past year, as defined in DSM-IV criteria. A history of schizophrenia (meeting DSM-IV criteria).
3. History of severe drug or alcohol abuse within the past year;
4. Any significant systemic illness or unstable medical condition that may make it difficult to comply with the protocol, such as severe autoimmune diseases or a history of cancer.
5. Have significant hearing, visual, or cognitive impairments, or are unable to participate in interviews in a meaningful way.

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective sleep indicators and clinical sleep-related scales | From enrollment to the end of treatment at 4 weeks

SECONDARY OUTCOMES:
Resting-state electroencephalogram, resting-state functional magnetic resonance imaging, blood biochemical indicators | From enrollment to the end of treatment at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China